CLINICAL TRIAL: NCT01585220
Title: A Randomized, Multi-center, Double Masked, Matched Pairs, Active-controlled Clinical Trial to Evaluate the Efficacy and Safety of Injection With Neuramis as Compared to Restylane® in Correction of Nasolabial Fold
Brief Title: Efficacy and Safety Study of Neuramis in Correction of Nasolabial Fold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT_PRT_NLF01
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Nasolabial Fold
Keywords: WSRS; GAIS; HA filler; filler

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuramis (Experimental)
  Interventions: Device: HA filler
- Restylane® (Active Comparator)
  Interventions: Device: HA filler

INTERVENTIONS:
Device: HA filler — The study device and comparator device will be intradermally injected to each left and right nasolabial fold according to the randomization.

SUMMARY:
This study design is a randomized, multi-center, double Masked, matched Pairs, active-controlled clinical trial. Subjects who voluntarily signed the informed consent and are judged to be eligible for this study will be intradermally injected both of study device and comparator device. Subjects will be randomized to receive injection of study device and comparator device on their each nasolabial fold. Efficacy is evaluated based on the change in Wrinkle Severity Rating Scale (WSRS) from baseline. Safety will be assessed based on 24 weeks follow up visits and subject diary which will be given to subjects during the first 2 weeks after the injection. Any uncomfortable things and adverse events will be investigated from subeject diary and follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 30 and 75
2. Subjects who wanting to correct his/her nasolabial fold and attaining grade 3 or 4 in the Wrinkle Severity Rating Scale(WSRS) of nasolabial fold
3. Subjects whose nasolabial folds are visually symmetric
4. Subjects who agreed to restrict any treatment for the wrinkle correction at the lower orbital rim area for the duration of the study
5. Subjects who can understand and comply with the instructions and all visit schedule
6. Subjects who voluntarily decided the participation of the study and signed the informed consent

Exclusion Criteria:

1. Subjects who had anti-coagulant therapy(excluding low-dose aspirin therapy(100mg, maximum 300mg/day dose)) within 2 weeks from the screening date
2. Subjects who had previous treatment at the lower orbital rim for wrinkle correction(e.g., face lift, soft tissue augmentation, medium depth peels, dermal photorejuvenation) within 6 months from screening date
3. Subjects who were treated calcium hydroxyapatite at the NLF area within a year from screening date
4. Subjects who had dermal augmentation permanent implants(e.g., silicone, Softform®) at the NLF area
5. Subjects who have a scar or skin lesion which can be affect to efficacy to the NLF area
6. Subjects who had anaphylaxis or severe combined allergy or allergy to lidocain or hyaluronic acid
7. Subjects who had a history of keloid formation or hypertrophic scar
8. Subjects who have a skin disorder or wound infection in the NLF area
9. Subjects who participated in other clinical trial within 30 days from screening date
10. The childbearing subjects who disagreed with medically acceptable contraception(e.g., condom, oral contraceptives continuing at least 3 months, contraceptives for injection or insertion, intrauterine contraceptive devices)
11. Pregnant or lactating subjects
12. Patients who are not eligible for this study at the medical discretion of the investigator

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2012-08-30 (Actual); Study Completion 2012-10-30 (Actual)

PRIMARY OUTCOMES:
WSRS | 24 weeks after the injection
  The change between baseline and 24 weeks WSRS evaluated by the investigator in charge of live assessment

SECONDARY OUTCOMES:
WSRS | 2, 8, 16, 24 weeks after the injection
  The change between baseline and 2, 8, 16, 24 week WSRS evaluated by the investigator in charge of photographic assessment
WSRS | 2, 8, 16 weeks after the injection
  The change between baseline and 2, 8, 16 week WSRS evaluated by the investigator in charge of live assessment
GAIS | 2, 8, 16, 24 weeks after the injection
  The rate of subjects whose GAIS, evaluated by the investigator in charge of live assessment, is 1 point or above after 2, 8, 16, 24 weeks from the injection
GAIS | 2, 8, 16, 24 weeks after the injection
  The rate of subjects whose GAIS, evaluated by the subjects him/herselves, is 1 point or above after 2, 8, 16, 24 weeks from the injection
WSRS | 2, 8, 16, 24 weeks after the injection
  The rate of subjects whose change of WSRS, evaluated by the investigator in charge of live assessment, is 1 point or above after 2, 8, 16, 24 weeks of the injection
WSRS | 2, 8, 16, 24 weeks after the injection
  The rate of subjects whose change of WSRS, evaluated by the investigator in charge of photographic assessment, is 1 pointe or above after 2, 8, 16, 24 weeks of the injection
Number of adverse events in subjects | Up to 24 weeks
  Adverse events occured after informed consent, Adverse drug events, Serious adverse events, lab test, physical examination, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Chan Yeong Heo, Principal Investigator — Seoul National University Bundang Hospital; Saik Bang, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Gangnam
  - Seoul National University Bundang Hospital, Seongnam, Gyunggi

REFERENCES:
- [Derived] Pak C, Park J, Hong J, Jeong J, Bang S, Heo CY. A Phase III, Randomized, Multi-Center, Double-Masked, Matched-Pairs, Active-Controlled Trial to Compare the Efficacy and Safety between Neuramis Deep and Restylane in the Correction of Nasolabial Folds. Arch Plast Surg. 2015 Nov;42(6):721-8. doi: 10.5999/aps.2015.42.6.721. Epub 2015 Nov 16. PMID 26618119